CLINICAL TRIAL: NCT00002383
Title: A Randomized, Parallel, Open-Label Study Comparing Saquinavir (Hard Gelatin Formulation, 600 Mg Tid) to Saquinavir Soft Gelatin Formulation [(400 Mg, 800 Mg, 1200 Mg) Tid} x 4 Weeks in HIV Infected Patients
Brief Title: A Comparison of Saquinavir Hard- and Soft-Gelatin Capsules in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 229M; NV15107
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-07

CONDITIONS: HIV Infections
Keywords: Drug Administration Schedule; HIV Protease Inhibitors; Dosage Forms; Saquinavir; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir

INTERVENTIONS:
Drug: Saquinavir

SUMMARY:
To compare the antiviral activity, safety, and pharmacokinetics of saquinavir hard gel capsule (HGC) formulation, to 1 of 3 doses of saquinavir soft gel capsule (SGC) formulation administered orally every 8 hours for 4 weeks.

DETAILED DESCRIPTION:
Patients are randomly assigned to one of the four treatment groups as follows:

Group 1: 10 patients receive saquinavir HGC. Group 2: 10 patients receive saquinavir SGC. Group 3: 30 patients receive saquinavir SGC at an intermediate dose. Group 4: 30 patients receive saquinavir SGC at the highest study dose. Upon completion of the initial 4 weeks, all patients may have the option to continue their originally-assigned therapy as monotherapy unless significant drug toxicity intervenes. If the analysis of the initial 4 week data identifies an optimal dose of saquinavir SGC, patients may have the option to change to this optimal dose in a treatment extension phase of the protocol. Patients in this extension phase may choose to remain on monotherapy unless they experience significant drug toxicity, their CD4 count or HIV-RNA levels return to baseline, until saquinavir is approved by the FDA or study termination, whichever comes first.

NOTE: A washout >= 28 days is required for patients on antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* CD4 count of 100 to 500 cells/mm3.
* Greater than 20,000 HIV-RNA copies/ml.

Exclusion Criteria

Prior Medication:

Excluded:

Prior treatment with protease inhibitors.

Required:

* Less than 8 weeks prior antiretroviral treatment (For at least 25% of patients).
* At least 8 weeks prior antiretroviral treatment (For at least 25% of patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Univ of Alabama at Birmingham / 1917 Rsch Cln, Birmingham, Alabama
  - Davis Med Ctr, San Francisco, California
  - Mt Zion Hosp of UCSF / HIV Research Ctr, San Francisco, California
  - Pacific Oaks Med Group / Research & Scientific Investiga, Sherman Oaks, California
  - Tulane Univ Med Ctr / Infectious Diseases Sect, New Orleans, Louisiana
  - New England Med Ctr, Boston, Massachusetts
  - Kansas City AIDS Research Consortium, Kansas City, Missouri
  - Harkness Pavilion, New York, New York
  - Oregon Health Sciences Univ, Portland, Oregon
  - Univ of Texas Med Branch / Virology Clinic, Galveston, Texas

REFERENCES:
- [Background] Cadman J. Roche brings new formulation of saquinavir to FDA. Food and Drug Administration. GMHC Treat Issues. 1997 Apr-May;11(4/5):8. PMID 11364377